CLINICAL TRIAL: NCT06974695
Title: Predictive Factors for Cholangioscopy-Assisted Lithotripsy Failure in the Management of Complex Biliary Stones: A Retrospective Analysis
Brief Title: Identification of Predictive Factors for Failure of Cholangioscopy-assisted Lithotripsy in the Management of Complex Bile Duct Stones: a Retrospective Study
Acronym: CLEVER
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Marion SCHAEFER, Hospital practitioner, Central Hospital, Nancy, France
Other Study IDs: 2025_PI_011
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Bile Duct Stones
Keywords: Cholangioscopy; Spyglass; Failure; Complex bile duct stone; predictive factor; electrohydraulic lithotripsy; EHL; lithotripsy; ERCP
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to optimize the management of complex biliary stones by identifying predictive factors for SpyGlass lithotripsy failure.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who underwent cholangioscopy-guided lithotripsy for bile duct stones between January 1, 2018, and May 30, 2025

Exclusion Criteria:

* Patient who objected to the collection of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient who underwent cholangioscopy-guided lithotripsy for bile duct stones between January 1, 2018, and May 30, 2025
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Predictive factors for failure of cholangioscopy lithotripsy in the management of complex bile duct stone | Baseline
  Cholangioscopy-guided lithotripsy failure: defined as stone clearance requiring more than one lithotripsy session or surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marion SCHAEFER, hospital practitioner, Study Director
Locations (1):
- CHRU Brabois Vandoeuvre les Nancy, Vandœuvre-lès-Nancy, Lorraine, France